CLINICAL TRIAL: NCT02918136
Title: Safety and Efficacy of Adult Adipose-Derived Stem Cell Injections Into Partial Thickness Rotator Cuff Tears
Brief Title: Safety and Efficacy Adipose-Derived Stem Cell Injection Partial Thickness Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InGeneron, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RTC-001
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Rotator Cuff Tear - Partial Thickness
MeSH Terms: interventions — Steroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- adipose-derived stem cell injection (Experimental): ultrasound guided injection of 5cc of adipose-derived stem cells (ADSCs)
  Interventions: Biological: Adipose derived regenerative cells
- cortisone injection (Active Comparator): ultrasound guided injection of cortisone
  Interventions: Drug: Cortisone Injectable

INTERVENTIONS:
Biological: Adipose derived regenerative cells
  Other Names: ADRCs
  Arms: adipose-derived stem cell injection
Drug: Cortisone Injectable
  Other Names: steroid
  Arms: cortisone injection

SUMMARY:
This is a prospective, randomized, multi-site, safety and efficacy study in subjects with rotator cuff injuries.

Patients will fall into two categories: treatment group (12 subjects) and non-treatment or control group (six subjects). The treatment group will undergo a small liposuction procedure and receive rotator cuff repair treatment with an ultrasound-guided injection of 5cc adipose-derived stem cells (ADSCs) into the point of injury. The control group will receive a 5cc cortisone injection into the point of injury

DETAILED DESCRIPTION:
The primary objectives of this study were to evaluate the safety of adult Adipose-Derived Stem Cell (ADRC) injection into partial thickness rotator cuff tears as indicated through adverse event rate and efficacy of pain and function through Rand short form-36 questionnaire and ASES Shoulder Score health questionnaires.

The secondary objective of this study was to assess the efficacy of adult ADRC injection into partial thickness rotator cuff tears through MRIs pre-and post-injection for the therapeutics intent to treat a rotator cuff injury.

Patients enrolled on this study received either ADRC (i.e., investigational treatment group) or TAU (i.e., control group). The investigational treatment group underwent a small liposuction procedure and received rotator cuff repair treatment with an ultrasound-guided injection of 5cc ADRCs into the point of injury. The control group received a 5cc cortisone injection. All patients, regardless of treatment, were followed up as indicated on the schedule of events table in the clinical study protocol.

Two clinical trial sites (Sioux Falls, SD and Fargo ND) enrolled subjects in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 30-75 years of age.
2. Clinical symptoms consistent with a rotator cuff lesion including but not limited to pain, muscle weakness, or active-limited range of motion (AROM).
3. Subjects who have not responded to physical therapy treatments for at least six weeks.
4. Subjects with > 70% passive range of motion (PROM).
5. Diagnosed with >50% tear to supraspinatus muscle or < 5mm separation assessed by MRI.
6. Diagnosed with a partial-thickness rotator cuff tear
7. The ability of subjects to give appropriate consent or have an appropriate representative available.

Exclusion Criteria:

1. Age <30 or > 75
2. Insufficient amount of subcutaneous tissue to allow recovery of 50cc of lipoaspirate.
3. History of systemic malignant neoplasms within last 5 years.
4. History of local neoplasm within the last 6 months and any history of local neoplasm at site of administration.
5. Subject is receiving immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.).
6. Subjects who are known to be HIV positive
7. Patients who have received a corticosteroid injection in rotator cuff site within last 3 months
8. Severe arthrosis of the glenohumeral or acromioclavicular joint
9. Irreparable rotator cuff tear (including rotator cuff tear arthropathy)
10. Fatty atrophy above Grade 2 in affected shoulder
11. Previous shoulder surgeries in affected shoulder
12. History of tobacco use within the last 3 months
13. Any contraindications to MRI scan according to MRI guidelines, or unwillingness to undergo MRI procedures
14. Patients on an active regimen of chemotherapy
15. Patients with a documented history of liver disease or an ALT value >400
16. Allergy to sodium citrate of any "caine" type of local anesthetic
17. Patients pregnant or breast feeding
18. Subject is in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason. This includes completion of Patient Reported Outcome instruments.
19. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
20. Subject is part of a vulnerable population who, in the judgment of the investigator, is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include: Individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.
21. Uncooperative patients or those with neurological/psychiatric disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-12; Primary Completion 2018-07-31 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
safety evaluation as indicated by collection of adverse events | enrollment through 12months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hurd, M.D., Principal Investigator — Sanford Orthopedics & Sports Medicine - Sioux Falls, SD
Locations (2):
- United States (2):
  - Sanford Orthopedics and Sports Medicine - Fargo, Fargo, North Dakota
  - Sanford orthopedics and Sports Medicine - Sioux Falls, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hurd JL, Facile TR, Weiss J, Hayes M, Hayes M, Furia JP, Maffulli N, Winnier GE, Alt C, Schmitz C, Alt EU, Lundeen M. Safety and efficacy of treating symptomatic, partial-thickness rotator cuff tears with fresh, uncultured, unmodified, autologous adipose-derived regenerative cells (UA-ADRCs) isolated at the point of care: a prospective, randomized, controlled first-in-human pilot study. J Orthop Surg Res. 2020 Mar 30;15(1):122. doi: 10.1186/s13018-020-01631-8. PMID 32238172